CLINICAL TRIAL: NCT02798549
Title: Hepatitis B Virus Particles-bound Human Proteins : Identification in Clinical Samples and Implication in the Viral Life Cycle
Brief Title: HBV Virions Bound Proteins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2013.809
Record Dates: First submitted 2016-05-30; First posted 2016-06-14 (Estimated); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Hepatitis B Virus Infection
Keywords: HBV; liver
MeSH Terms: conditions — Hepatitis B | interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Viraemic (Other)
  Interventions: Other: blood draw
- Remission (Other)
  Interventions: Other: blood draw

INTERVENTIONS:
Other: blood draw — blood draw of 150ml, twice

SUMMARY:
The emergence of hepatocellular carcinoma (HCC) has prompted a search for a thorough understanding of the biology of one of its major causative agents, the hepatitis B virus (HBV). HBV particles acquire via budding and encapsidation cellular proteins. There is mounting evidence on several viral species that virion-bound proteins are prone to be involved either at the replication, budding/egress or entry/release steps of the viral cycle.

Identifying such targets may yield ideal candidates for gaining insight on the dependence of HBV upon a restricted subset of host proteins, therefore providing refined sets of genetically stable targets for therapy. This project's goals are to set up adequate conditions for robust and reproducible purification of HBV virions in clinical samples, followed by the identification of their HBV-bound host proteins and the characterization of their functions. Proteomics profiling of HBV particles purified from clinical samples will be overlaid with proteins identified and characterized in cell culture grown HBV particles, using clinical biomarker discovery grade criteria. Targets identified in both samples sets will be subjected to in vitro investigations using HBV-replicating cells. Conventional biochemical and imaging methods will be used in order to: (i) ascertain their physical association with HBV virions; (ii) define the modalities of their interaction with HBV proteins; (iii) decipher the topology and subcellular localization of their association with HBV proteins and virions; (iv) quantitatively assess their functional involvement in particle budding, egress or secretion and infectivity. A candidate that yielded satisfactory results in these experiments will be disclosed and further investigated at the level of structural biology, in collaborative research programs.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria
* Adult> 18 and <60 years
* Infected with HBV.
* positive viremia for more than 6 months
* Viremia> 106 IU / ml.
* Immunotolerant individuals, untreated
* Aviraemic individuals,

Exclusion Criteria:

* patient with against-indication for a blood sample of 150 ml
* immunosuppressive therapy patient
* Patient with liver disease other than hepatitis B.
* patient with hepatocellular carcinoma.
* Patients with one or more severe co-morbidities defined as:
* Co-infection with HIV or hepatitis C virus (HCV).
* hematological malignancies changing or aplasia
* Insulin-dependent diabetes
* dialyzed chronic renal failure
* Heart failure
* Persons subject to legal protection or the subject of a safeguard measure of justice
* not affiliated with a social security scheme or not beneficiaries of such a scheme
* Pregnant women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2015-01-12 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Presence of a virion-bound protein identified by mass spectrometry | One to two years after mass spectrometry identification of the candidate

SECONDARY OUTCOMES:
Comparison of clinical virions datasets with in vitro grown virions datasets (mass spectrometry) | One to two years after mass spectrometry identification of the candidate
  Proteins identified from viral particles purified from clinical samples will be compared to proteins identified in viral particles from cells of human hepatocarcinoma origin.

CONTACTS AND LOCATIONS:
Overall Officials: Fabien Zoulim, Prof, Principal Investigator — Hospices Civils de Lyon, Univ. of Lyon, Inserm
Locations (1):
- Service d'Hépato-Gastroentérologie, Hopital de la Croix-Rousse, Hospices Civils de Lyon, Lyon, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cottarel J, Plissonnier ML, Kullolli M, Pitteri S, Clement S, Millarte V, Si-Ahmed SN, Farhan H, Zoulim F, Parent R. FIG4 is a hepatitis C virus particle-bound protein implicated in virion morphogenesis and infectivity with cholesteryl ester modulation potential. J Gen Virol. 2016 Jan;97(1):69-81. doi: 10.1099/jgv.0.000331. Epub 2015 Oct 29. PMID 26519381